CLINICAL TRIAL: NCT01404702
Title: Pilot Study of Zoledronic Acid and Interleukin-2 for Refractory Pediatric Neuroblastoma: Assessment of Tolerability and In Vivo Expansion γδ T-Cells
Brief Title: Pilot Study of Zoledronic Acid and Interleukin-2 for Refractory Pediatric Neuroblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Accrual slower than anticipated
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1051; F101013003 (Other: UAB Institutional Board for Human Use)
Record Dates: First submitted 2011-07-13; First posted 2011-07-28 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Pediatrics; Refractory; Immunotherapy; Biological therapy; Lymphocytes; Cancer; Bisphosphonate
MeSH Terms: conditions — Neuroblastoma; Neoplasms | interventions — Zoledronic Acid; aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zoledronic Acid and Interleukin-2 (Experimental)
  Interventions: Drug: Zoledronic Acid; Biological: Aldesleukin

INTERVENTIONS:
Drug: Zoledronic Acid — 4 mg/m2/dose given iv on day 0 of every 28 day cycle
  Other Names: Zometa
Biological: Aldesleukin — Dose Level 1: 3 x 10^6 IU/m2/day given subcutaneously on days 0 through 4 and 14 through 18 every 28 day cycle
  Dose Level 2: 6 x 10^6 IU/m2/day given subcutaneously on days 0 through 4 and 14 through 18 every 28 day cycle
  Other Names: Proleukin; Interleukin-2

SUMMARY:
Neuroblastoma (NB) is the most common extracranial solid tumor in children, with an annual incidence of 10.5 per million children less than 15 years of age. NB accounts for 15% of childhood cancer deaths. High risk (HR) patients carry a poor prognosis despite treatment with intensive chemotherapy, surgery and/or radiation, autologous bone marrow transplant, and treatment with cis-retinoic acid. New therapies are desperately needed for such patients. Recently, it has been demonstrated that HR NB patients benefit from anti-GD2 antibody therapy which directs the immune system against NB cells. To further explore means of harnessing the immune system to attack NB, the investigators are studying the combination of zoledronic acid (ZOL) and interleukin-2 (IL-2). ZOL has been demonstrated to have direct anti-neuroblastoma effects in laboratory studies. ZOL also augments the production of tumor killing white blood cells called gamma-delta T cells. When used in combination with IL-2, ZOL is capable of eliciting potent anti-cancer effects in patients, in part, via the expansion of gamma-delta T cells. In this present trial the investigators aim to study the tolerability of the combination of ZOL and IL-2 in pediatric NB patients. Patients will also be monitored radiologically for tumor response to therapy. Correlative biological studies will study the ability of this drug combination to elicit the production of NB killing gamma-delta T cells in children.

ELIGIBILITY:
Inclusion Criteria:

* All patients must be diagnosed with treatment-refractory neuroblastoma with no known curative treatment options. Tumor histology should be verified at diagnosis or relapse.
* Prior to enrollment, a determination of residual disease must be performed
* Patients must have a Lansky or Karnofsky performance scale score of ≥ 50%.
* Patients must have a life expectancy of ≥ 2 months (8 weeks).
* Total absolute neutrophil count (ANC) is at least 750, Hgb≥8 grams/dl, and plts ≥ 75K. PRBC transfusions are allowed.
* Patients with bone marrow disease will not evaluable for hematologic toxicity. These patients must have a peripheral absolute neutrophil count

  * 750, platelet count ≥ 50K and Hgb ≥8 grams/dl. Transfusions are permitted to meet both the platelet and hemoglobin criteria.
* Creatinine clearance or radioisotope GFR > 70mL/min/1.73 m2 or a serum creatinine based on age/gender as follows:
* ≤ 0.8 mg/dL (for patients 2 to 5 years of age)
* ≤ 1.0 mg/dL (for patients 6 to 9 years of age)
* ≤ 1.2 mg/dL (for patients 10 to 12 years of age)
* ≤ 1.4 mg/dL (for female patients ≥ 13 years of age)
* ≤ 1.5 mg/dL (for male patients 13 to 15 years of age)
* ≤ 1.6 mg/dL (for male patients ≥ 16 years of age)
* Total bilirubin ≤ 2.5 x upper limit of normal (ULN) for age, and
* SGPT (ALT) < 2.5 x upper limit of normal (ULN) for age.
* SOS (sinusoidal obstruction syndrome, formerly known as veno-occlusive disease [VOD]), if present, should be stable or improving.
* Shortening fraction of > 27% by echocardiogram, or ejection fraction of > 55% by radionuclide angiography.
* No evidence of dyspnea at rest. If PFTs are performed, FEV1/FVC > 60% by pulmonary function test.
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled.
* CNS toxicity < Grade 2.

Exclusion Criteria:

* Females of childbearing potential must have a negative pregnancy test.
* Patients of childbearing potential must agree to use an effective birth control method.
* Female patients who are lactating must agree to stop breast-feeding.
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional requirements for human studies must be met.
* Previous treatment with anti-GD2 and interleukin2 therapy

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and toxicity of zoledronic acid and aldesleukin | 1.5 years
  The NCI Common Terminology Criteria for AEs will be used for reporting & identification of dose limiting toxicities. DLTs will include any grade 3 non-hematologic toxicity not included here: Gr 3 nausea & vomiting & diarrhea, Gr 3 fever, Gr 3 skin toxicity that remains stable & tolerable, or improves with treatment within 24 hrs, Gr 3 neurotoxicity with subjective findings, Gr 4 hematologic toxicity, which improves to at least Gr 2 or baseline pre-therapy values within one week of completing IL2 infusion, Gr 3 performance that returns to 50 or higher before the start of the next therapy cycle.

SECONDARY OUTCOMES:
Evaluate the biologic function of autologous expanded/activated gamma delta T cells in neuroblastoma patients receiving therapy with zoledronic acid and aldesleukin | 3 years
  The ability of gamma-delta T cells derived from patients' peripheral blood to kill NB cells in vitro will be quantified by standard tumor cytotoxicity assays.
Evaluate immune phenotype of in vivo expanded/activated autologous gamma delta T cells | 3 years
  Peripheral blood mononuclear cells will be immunophenotyped by standard conjugation of fluorescent monoclonal antibodies in order to quantify and phenotype patient lymphocytes using flow cytometry.
To document tumor response in patients with measurable disease. | 3 years
  Tumor response and progression will be assessed and documented utilizing the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
Determine the ability of in vivo expanded/activated gamma delta T cells to infiltrate neuroblastoma tissue using immunohistochemical techniques when post-therapy specimens are available. | 3 years
  Patients with known or suspected bone marrow metastasis will undergo bilateral bone marrow biopsies at the beginning and end of the first course of therapy. This tissue will be fixed and processed per protocol (Appendix I) and infiltrating lymphocytes per hpf will be documented under standard microscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Pressey, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham-Children's of Alabama, Birmingham, Alabama, United States